CLINICAL TRIAL: NCT05761158
Title: Study of the Characteristics of Pruritus in Patients With Frontal Fibrosing Alopecia or Lichen Planus Pilaris
Acronym: PRURIT-ALOPECI
Status: Terminated | Type: Observational
Why Stopped: Discontinuation of the study was justified by the inclusion of 21/100 patients, which finally enabled a relevant analysis to be made in view of the homogeneity of the results.
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0227
Record Dates: First submitted 2023-02-01; First posted 2023-03-09 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-01

CONDITIONS: Alopecia; Lichen Planus
MeSH Terms: conditions — Alopecia; Lichen Planus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: patients answer the same questionnaire whether they have frontal alopecia or lichen planus pilaris
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — patients are asked to complete a questionnaire

SUMMARY:
The prevalence of pruritus has been studied in frontal fibrosis alopecia (FFA) and lichen planus pilaris (LPP), but there are no studies evaluating the characteristics of pruritus, the correlation between pruritus and disease activity, and its impact on quality of life.

The knowledge of the characteristics of pruritus, of the link "disease activity - pruritus", and its impact on the quality of life could allow us to modify the management of the patient (modification or intensification of therapy, close monitoring...)

ELIGIBILITY:
Inclusion Criteria:

* Major patient.
* Fibrosing frontal alopecia or lichen planus pilaris
* Presence of pruritus of the scalp : a positive response to the question "do you experience itchy scalp?"
* The patient received an information note and did not object to the study

Exclusion Criteria:

* Patients under 18 years of age.
* Other pathologies causing scalp pruritus (seborrheic dermatitis, contact dermatitis, lupus, Quinquaud's decalcifying folliculitis, ectoparasitosis, scalp psoriasis, ringworm, red sclap syndrome, dermatomyositis, central centrifugal cicatricial alopecia (CCCA))
* Refusal to participate by the patient.
* Patient under legal protection (curatorship, guardianship, ...)
* Patient not covered by social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients with frontal fibrosing alopecia or lichen planus pilaris, with scalp pruritus, followed in the Dermatology Department of the CHRU Brest and having given their consent to participate in the study.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Study of the characteristics of pruritus in patients with frontal fibrosis alopecia or lichen planus pilaris | Hour1
  Questionnaire of Brest
Study of the characteristics of pruritus in patients with frontal fibrosis alopecia or lichen | Hour1
  5D itch scale

SECONDARY OUTCOMES:
Study the relationship between disease activity (AFF or LPP) and pruritus, as well as the impact of pruritus on patients' quality of life. | Hour1
  ItchyQol (Itchy Quality of Life)
Study the relationship between disease activity (AFF or LPP) and pruritus, as well as the impact of pruritus on patients' quality of life. | Hour1
  Questionnaire of FFASI
Study the relationship between disease activity (AFF or LPP) and pruritus, as well as the impact of pruritus on patients' quality of life. | Hour1
  Questionnaire of LPPAI

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.